CLINICAL TRIAL: NCT04823364
Title: Measuring Glutamate and GABA Brain Levels in Adults With Attention Deficit Hyperactivity Disorder (ADHD) Using Magnetic Resonance Spectroscopy (MRS)
Brief Title: Evaluation of Brain Neurotransmitter Levels in Adults With ADHD, Before and After Stimulant Treatment
Acronym: ADHD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Professor Assaf Tal left Weizmann Institute
Sponsor: Weizmann Institute of Science (Other)
Collaborators: Tel Aviv University (Other); Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0109-19-MOH
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2022-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ACC; methylphenidate; MRS; Glutamate; GABA
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Group 1 control healthy people Group 2 ADHD
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Medically healthy adults diagnosed with ADHD (Active Comparator): Medically healthy adults diagnosed with ADHD (men and women) ages 18-40 years (N= 35), treated with Amphetamines (Mixed Amphetamine salts (Attent) or short-acting methylphenidate (Ritalin)
  Interventions: Other: Neurotransmitters evaluation by MRS
- Control (No Intervention): HCS (N= 25) volunteers ages 18-40 years, who did not report ADHD or any other illness or medical conditions, and who do not take chronically medications, will be enrolled from the general population.

INTERVENTIONS:
Other: Neurotransmitters evaluation by MRS — Baseline MRS screening for volunteers and ADHD groups and repeated measurement for ADHD group after taking stimulant drug treatment
  Arms: Medically healthy adults diagnosed with ADHD

SUMMARY:
Background:

Attention deficit hyperactivity disorder (ADHD) is one of the most prevalent neurobiological brain disorders. Diagnosis of ADHD in adults is complex and subjective. Recent studies give further support for the involvement of glutamatergic and GABAergic neurotransmitters in the pathophysiology of ADHD. Studies show that glutamate (Glu) and GABA change according to stimulant treatment. Measuring modulations in the anterior cingulate cortex (ACC) of Glu and GABA may help to explore the pathophysiology of ADHD and give a diagnostic biomarker tool for ADHD in adults.

Aim:

To characterize Glu and GABA levels in the ACC, by using the proton Magnetic Resonance Spectroscopy ([1H]MRS) system in adults with ADHD compared to healthy control subjects (HCS), before and after stimulant treatment, and to correlate between Glu and GABA levels and clinical symptoms.

Method:

ADHD adults ages 18-40 years (N= 35), and HCS (N= 25), will fill out a DSMV and ASRS questionnaire.

Spectroscopic analyses will be done using 1H MRS (3T) in ADHD adults, before and after stimulant treatment (Methylphenidate /Mixed Amphetamine salts) in an open-label fashion as compared to HCS. Proton spectra will be acquired from the ACC.

DETAILED DESCRIPTION:
Hypothesis:

1. We hypothesize that brain Glu and GABA levels and/or their ratio involved in ADHD pathology
2. Glu and GABA levels and/or their ratio will be affected by medical treatment in ADHD group
3. Alteration of Glu and GABA and/or their ratios, before and after treatment, will correlate with clinical response to treatment

Primary Objectives:

To characterize changes in Glu and GABA levels in the ACC of adults with ADHD compared to the healthy subjects To characterize Glu and GABA levels in the ACC of adults with ADHD before and 1.5 hrs. after stimulant treatment using 1H MRS system.

Secondary objective:

To study the correlation between Glu and GABA levels in ADHD patients (before and after medical treatment) and clinical symptoms as assessed by ASRS and DSMV and/or NeuroTrax Braincare computerized test

Design and study population:

This is a prospective observational, open-label, comparative study that is approved by the Institutional Review Board (IRB) of Maccabi Healthcare services and the Ethical Committee of Tel Aviv University, in collaboration with the Weizmann Institute of Science. Medically healthy ADHD adults of ages 18-40 years (N= 35), and matched HCS (N= 25) will be recruited.

Procedure ADHD Participants will be enrolled from the Maccabi database. Volunteers will be enrolled as a Control group

* Pre-assessment questionnaires including epidemiologic data, DSMV, and Adult ADHD Self-Report Scale (ASRS) will be filled out.
* Detailed explanation will be given of the trial objectives, trial methods and risks or possible discomfort that may result from an MRI/MRS examination
* During screening, subjects will receive information regarding the study, including general eligibility criteria, study design, procedures and duration. Subjects will have the opportunity to ask questions and will undergo an informed consent procedure. Subjects meeting inclusion/exclusion criteria will be enrolled. The participant will sign an informed consent form and will receive a copy.

After screening, participants who meet the inclusion criteria will be invited to the center for Computational Neuroimaging at Weizmann Institute of Science to perform the MRS scan.

ADHD patients will be instructed not to take medication for at least 72 hours prior to their arrival and will be asked to bring their medical drug treatment.

All participants will go through spectroscopic analyses using 1H MRS (at 3 Tesla) Control group participants will go through MRS once and complete their study. Adults with ADHD will repeat MRS screening, 1.5 hours after taking their medical treatment (Methylphenidate /Mixed Amphetamine salts).

Study population:

Medically healthy adults diagnosed with ADHD (men and women) ages 18-40 years (N= 35), treated with Amphetamines (Mixed Amphetamine salts (Attent) or short-acting methylphenidate (Ritalin)) will be enrolled from the Maccabi database. Matched HCS (N= 25) volunteers ages 18-40 years, who did not report ADHD or any other illness or medical conditions, and who do not take chronic medications, will be enrolled from the general population.

The Adult ADHD Self-Report Scale and DSMV questionnaire will be used to determine ADHD symptoms in both groups.

ELIGIBILITY:
Inclusion Criteria:

Giving informed written consent to participate on a voluntary basis.

For the healthy control group:

Men and women aged 18-40 years, who did not report ADHD or any other chronic or psychiatric illness or medical conditions (at most two symptoms of inattention and/or hyperactivity/impulsivity).

For the ADHD group patients:

1. Men and women aged 18-40 years, who have a diagnosis of ADHD, according to DSM V criteria by a Neurologist.
2. Have a valid prescription for Mixed Amphetamine salts (Attent) or short-acting methylphenidate (Ritalin) for ADHD
3. Withhold medication 72h prior to MRS scan.

Exclusion Criteria:

Exclusion criteria identical for patients and control group:

1. Subjects with metallic devices that precludemagnetic resonance imaging or any silver part that is not MRI compliant
2. Current presence of any other DSM V psychiatric disorder
3. Significant medical or neurological illness affecting brain function
4. Subjects with any clinically signiﬁcant or unstable medical conditions
5. Use of any psychotropic medication, other than stimulants, in the previous 3 months
6. Pregnant women
7. BMI > 35
8. History of brain MRI
9. A patient who does not agree that the scan will be decoded by a radiologist
10. A patient who does not agree that in case of an abnormal finding, the imaging results will be forwarded to the attending physician for further clarification
11. Understanding and/or language problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Glu and GABA levels measured by MRS in ACC brain area | 72 hours without stimulant
  Differences in levels of Glu and GABA in ADHD patients compared to healthy volunteers
Glu and GABA levels measured by MRS in ACC brain area before and after medical treatment | 90 minutes after stimulant
  Differences in levels of Glu and GABA measured before and after medical treatment.

SECONDARY OUTCOMES:
Correlation of Glu and GABA levels with clinical symptoms before and after stimulants | 210 minutes after stimulant
  Analysis of correlation of Glu and GABA levels with post/previous clinical manifestation evaluated by Neuro Trax Braincare test and/or ASRS and DSMV questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Tal, PhD., Study Chair — Maccabi Healthcare Services, Israel
Locations (2):
- Israel (2):
  - Maccabi Health Services, Kfar Saba
  - Weizmann, Rehovot

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data generated by this project is an essential part of our proposed activities and will be carried out in several different ways. We would wish to make our results available both to the community of scientists interested in ADHD and the biology to avoid unintentional duplication of research. Conversely, we would welcome collaboration with others who could make use of the H-MRS protocols developed in psychiatric disease. Any patient-level data that is shared will be anonymized to protect personally identifiable information.
Supporting Information: Study Protocol
Time Frame: 4 years
Access Criteria: Broad sharing of the data will be communicated through NDA and its support staff according to the Provisions for Data Submission and Data Sharing Schedule. The findings of this research will be de-identified data, such that the identities of participants cannot be readily ascertained or otherwise associated with the data by NDA staff or secondary data users.

REFERENCES:
- [Background] Naaijen J, Lythgoe DJ, Amiri H, Buitelaar JK, Glennon JC. Fronto-striatal glutamatergic compounds in compulsive and impulsive syndromes: a review of magnetic resonance spectroscopy studies. Neurosci Biobehav Rev. 2015 May;52:74-88. doi: 10.1016/j.neubiorev.2015.02.009. Epub 2015 Feb 21. PMID 25712432
- [Background] Maltezos S, Horder J, Coghlan S, Skirrow C, O'Gorman R, Lavender TJ, Mendez MA, Mehta M, Daly E, Xenitidis K, Paliokosta E, Spain D, Pitts M, Asherson P, Lythgoe DJ, Barker GJ, Murphy DG. Glutamate/glutamine and neuronal integrity in adults with ADHD: a proton MRS study. Transl Psychiatry. 2014 Mar 18;4(3):e373. doi: 10.1038/tp.2014.11. PMID 24643164
- [Background] Ende G, Cackowski S, Van Eijk J, Sack M, Demirakca T, Kleindienst N, Bohus M, Sobanski E, Krause-Utz A, Schmahl C. Impulsivity and Aggression in Female BPD and ADHD Patients: Association with ACC Glutamate and GABA Concentrations. Neuropsychopharmacology. 2016 Jan;41(2):410-8. doi: 10.1038/npp.2015.153. Epub 2015 Jun 4. PMID 26040503
- [Background] Bauer J, Werner A, Kohl W, Kugel H, Shushakova A, Pedersen A, Ohrmann P. Hyperactivity and impulsivity in adult attention-deficit/hyperactivity disorder is related to glutamatergic dysfunction in the anterior cingulate cortex. World J Biol Psychiatry. 2018 Oct;19(7):538-546. doi: 10.1080/15622975.2016.1262060. Epub 2016 Dec 15. PMID 27973969
- [Background] Perlov E, Philipsen A, Hesslinger B, Buechert M, Ahrendts J, Feige B, Bubl E, Hennig J, Ebert D, Tebartz van Elst L. Reduced cingulate glutamate/glutamine-to-creatine ratios in adult patients with attention deficit/hyperactivity disorder -- a magnet resonance spectroscopy study. J Psychiatr Res. 2007 Dec;41(11):934-41. doi: 10.1016/j.jpsychires.2006.12.007. Epub 2007 Feb 15. PMID 17303167
- [Background] Endres D, Perlov E, Maier S, Feige B, Nickel K, Goll P, Bubl E, Lange T, Glauche V, Graf E, Ebert D, Sobanski E, Philipsen A, Tebartz van Elst L. Normal Neurochemistry in the Prefrontal and Cerebellar Brain of Adults with Attention-Deficit Hyperactivity Disorder. Front Behav Neurosci. 2015 Sep 28;9:242. doi: 10.3389/fnbeh.2015.00242. eCollection 2015. PMID 26441572
- [Background] Bezalel V, Paz R, Tal A. Inhibitory and excitatory mechanisms in the human cingulate-cortex support reinforcement learning: A functional Proton Magnetic Resonance Spectroscopy study. Neuroimage. 2019 Jan 1;184:25-35. doi: 10.1016/j.neuroimage.2018.09.016. Epub 2018 Sep 7. PMID 30201464